CLINICAL TRIAL: NCT05254015
Title: Cognitive Rehabilitation and Exposure Therapy for Geriatric Hoarding
Acronym: CREST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Catherine Ayers, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01MH127056-01A1 (NIH)
Record Dates: First submitted 2022-02-09; First posted 2022-02-24 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Hoarding Disorder; Obsessive-Compulsive Disorder
Keywords: older adult; executive dysfunction; hoarding; OCD; exposure therapy; cognitive rehabilitation
MeSH Terms: conditions — Hoarding Disorder; Obsessive-Compulsive Disorder; Hoarding | interventions — Cognitive Training; Case Management

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Rehabilitation and Exposure/Sorting Therapy (CREST) (Experimental): Compensatory Cognitive Training (CCT) Modules (7 sessions). Compensatory Cognitive Training is a manualized, low-tech, cognitive training intervention designed to target cognitive impairments common in people with psychiatric illnesses. The CCT modules specifically selected for CREST map onto known areas of HD neurocognitive impairments and include training in prospective memory, prioritizing, problem solving, planning, and cognitive flexibility.
  Exposure to Discarding and Acquiring Modules (19 sessions). Symptoms of acquiring and saving are themselves avoidance behaviors to avoid internal distress related to negative thoughts and emotions. ET utilizes in vivo exposure exercises taking place in the home to enhance generalization of their new skills. Fear hierarchies typically start with a space that has low clutter volume or there is less of an urge to save a particular type of item in that environment.
  Interventions: Behavioral: Cognitive Rehabilitation and Exposure/Sorting Therapy (CREST)
- Case Management (CM) (Active Comparator): Case Management (CM). CM consists of a set of well-established strategies commonly used in community service settings to address serious and complex problems in particularly vulnerable and often marginalized populations such as those with HD.
  Interventions: Behavioral: Case Management

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation and Exposure/Sorting Therapy (CREST) — Cognitive Rehabilitation and Exposure/Sorting Therapy (CREST) includes cognitive rehabilitation of executive functioning and exposure therapy for discarding/not acquiring.
  Arms: Cognitive Rehabilitation and Exposure/Sorting Therapy (CREST)
Behavioral: Case Management — Case management includes linking to resources, monitoring health, and safety hazards.
  Arms: Case Management (CM)

SUMMARY:
Hoarding disorder (HD) is a chronic, progressive, and debilitating psychiatric condition that leads to devastating personal and public consequences, particularly for older adults. This confirmatory efficacy trial will advance our knowledge of the mechanisms of action in the treatment of HD as well as reduce symptom severity, disability, and community consequences.

DETAILED DESCRIPTION:
Hoarding disorder (HD) is a chronic, progressive, and debilitating psychiatric condition that leads to devastating personal and community consequences, particularly for older adults. HD is defined by persistent difficulty discarding or parting with possessions due to distress associated with discarding, urges to save, and/or difficulty making decisions about what to keep and what to discard. As a result, clutter accumulates and fills active living areas, preventing the normal use of space and resulting in distress and disability. Community epidemiological reports estimate the prevalence of clinically significant hoarding symptoms at 7% in individuals over age 60 and even higher rates in those over age 70. HD is the only neuropsychiatric condition that progresses in severity and population prevalence with age apart from dementia.

Inhibition and cognitive switching have been identified as key deficits in older adults with HD. These executive functioning areas are consistent with the RDoC cognitive control domain and particularly the goal selection, updating, representation, and maintenance subconstruct. Findings suggest that these deficits may contribute to the symptomatic expression of HD, degree of functional impairment, and modest responses to HD treatment. Furthermore, anticipatory and experiential fear and anxiety, consistent with the RDoC constructs of acute and potential threat, lead to sustained problems with discarding items and clutter accumulation. When these constructs are targeted, our group has produced clinically and statistically significant outcomes.

Consistent with NIMH strategic goal 3.1, to arrive at effective treatment approaches for unmet therapeutic domains in behavioral science, this project seeks to conduct the first confirmatory efficacy trial for older adults with HD. We propose a RCT comparing CREST to a case management control condition for 150 adults age 50 and older with HD. We are examining age as a moderator and will therefore include both midlife and late life participants. An evaluation of treatment outcome, including hoarding severity and functional outcomes, will be conducted at baseline (0 months), mid-treatment (3 months), end of treatment (6 months), 3-month (9 months) and 6-month follow-up (12 months). Participants will receive 26 weekly 60-minute individual sessions over the course of 32 weeks maximum (6-7.5 months). They will receive 50% in home and 50% office visits. We will examine factors that mediate improvement in CREST (improved inhibition/cognitive switching and reduction in fear/anxiety of discarding items) through physiological, behavioral, self-report, and paradigm assessments. Individual factors (e.g., age and other demographic factors, baseline cognitive control, baseline hoarding severity) and treatment factors (e.g., session attendance) will be evaluated as moderators. The specific aims include determining confirmatory efficacy of CREST, mechanisms of CREST effects, and moderators of CREST. If successful, this project would lead to an effectiveness trial in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

* adults age 50 and older
* voluntary informed consent for participation
* DSM-5 diagnosis of HD
* HD as a primary, most severe diagnosis
* stable on medications for at least 8 weeks

Exclusion Criteria:

* current psychosis or mania as measured by the Mini-International
* current or history of any neurodegenerative disease
* substance use disorder
* current use of benzodiazepine medication
* suicidality
* current participation in exposure-based therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Saving Inventory-Revised (SI-R) | through study completion, an average of 1 year
  Hoarding symptom severity will be measured using the Saving Inventory-Revised (SI-R), a 23-item self-report measure used to assess common HD symptoms. Subscales include excessive clutter, compulsive acquisition, and difficulty discarding. The SI-R has demonstrated good internal consistency, concurrent validity, divergent validity, and test-retest reliability in clinical samples with HD. The total score will be used for analyses.
Change in Self-report Clutter Image Rating (CIR) | through study completion, an average of 1 year
  The Clutter Image Rating Scale (CIR) is a measure using a series of 9 photographs each of a kitchen, living room, and bedroom with varying levels of clutter. Participants and the rater independently select the photograph that most closely resembles each of the three rooms in the home. Internal consistency, test-retest reliability, inter-rater reliability, and correlations with validated HD measures for the CIR were high.

SECONDARY OUTCOMES:
PROMIS-43 Profile v2. | through study completion, an average of 1 year
  Functioning will be assessed with the PROMIS-43 Profile v2., which consists of a fixed collection of 6-item sets to assess global health and functioning (in physical, mental, and social domains). The PROMIS-43 assesses anxiety, depression, fatigue, pain interference, pain intensity, physical functioning, sleep disturbance, and ability to participate in social roles and activities. Substantial evidence supports the validity, reliability, and responsiveness to change of the PROMIS measures among adults with and without medical and mental health conditions.
UCSD Performance-Based Skills Assessment (UPSA-2) | through study completion, an average of 1 year
  The UCSD Performance-Based Skills Assessment (UPSA-2) is an assessment of everyday functioning skills involved in household management (e.g., writing a shopping list based on a provided recipe), communication (e.g., rescheduling a doctor's appointment), finance (e.g., paying a utility bill), comprehension/planning (e.g., planning an outing), medication management (taking medications as planned), and transportation (e.g., reading comprehension of a bus schedule). The UPSA-2 has demonstrated high inter-rater reliability (0.91) and convergent validity with other performance-based measures. The total UPSA-2 summary score will be used for analyses.
UCSD SORT Test (U-SORT) | through study completion, an average of 1 year
  The UCSD SORT Test (U-SORT) will be used to measure participants' organizational skills as they relate to functional capacity. During the administration of the U-SORT, participants are instructed to sort 42 household objects (e.g., bent and unbent paper clips, used and unused condiment packets) from a hypothetical "junk drawer" into either "keep" or "trash" piles. Participants are given two minutes to complete the task and one point is awarded for each correctly sorted item, for a total of 42 points. The U-SORT has high internal consistency (alpha = .86) and adequate convergent validity. The total U-SORT score will be used in analyses.

OTHER OUTCOMES:
DKEFS | through study completion, an average of 1 year
  Cognitive Control (inhibition and cognitive switching) will be assessed using the Delis-Kaplan Executive Function System (D-KEFS), which was specifically designed to detect deficits in high-level cognitive functions and has demonstrated strong reliability and validity in various clinical populations. We will administer five tests from the D-KEFS that examine components of executive functioning, including inhibition (the Color-Word Interference Test), cognitive switching (Verbal Fluency, Trails, Design Fluency), and Planning (Tower).
Behavior Rating Inventory of Executive Function- Adult Version (BRIEF-A) | through study completion, an average of 1 year
  The Behavior Rating Inventory of Executive Function- Adult Version (BRIEF-A) is a validated measure that captures views of an adult's executive functions or self-regulation their everyday environment. This will be used to assess nine non-overlapping theoretically and empirically derived clinical scales: Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organization.
Behavioral Avoidance Task (BAT) | through study completion, an average of 1 year
  Threat: Fear/Anxiety will be assessed via a Behavioral Avoidance Task (BAT), utilized for assessing avoidance to sorting and discarding possessions. The BAT has been validated for measuring avoidance in OCD samples, and will be adjusted for use in HD samples.
Heart Rate (HR) | through study completion, an average of 1 year
  Threat response to discarding in beats per minute during BAT.
Skin Conductance Response (SCR) | through study completion, an average of 1 year
  Threat response to discarding in changes in temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ayers, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Guava Hall, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this project includes self-report, observational, paradigm and physiology de-identified data from participants with hoarding disorder. During consent, participants will be provided with information about how their data will be shared. All de-identified data from this project will be shared in accordance with NIMH guidance via the NIMH Data Archive (NDA).
  Data will be individualized data of 150 participants. There will be no specialized tools or software that is required for access. Supporting documentation such as data collection instruments, protocols, data dictionaries and definitions will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared as soon as possible, and no later than time of an associated publication or end of a performance period. We will make data available for as long as we believe it could be useful to the scientific community.
Access Criteria: We will be using NDA and following the policies and procedures for access consistent with NIMH data policies. Access to databases generated under the project will be available for educational, research and non-profit purposes for non-commercial use. Such access will be provided using web-based applications and in a commonly used format.